CLINICAL TRIAL: NCT06756750
Title: Intraoperative Low-dose Glucocorticoids in Surgical Patients With Abdominal Sepsis: A Multicenter Retrospective Cohort Study
Brief Title: Clinical Characteristics and Risk Factors for In-Hospital Mortality in Surgical Patients With Abdominal Sepsis
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Professor, Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-L06
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Glucocorticoid
Keywords: abdominal sepsis; surgical patients; risk factors; general anesthesia; retrospective
MeSH Terms: conditions — Sepsis; Intraabdominal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study of sepsis patients with abdominal infections who underwent abdominal surgery was conducted in an attempt to reveal the epidemiological characteristics of sepsis after abdominal surgery, risk factors, and to analyze the prognosis of the patients, to reveal indicators of predictive value for the prognosis of patients with sepsis, with a view to providing certain evidence for optimizing the perianesthesia management of patients with sepsis.

DETAILED DESCRIPTION:
Background and Aims: Abdominal sepsis refers to a severe and potentially life-threatening condition characterized by the presence of infection, inflammation, and tissue damage within the abdominal cavity. Glucocorticoids (GCs) play an important role in regulation of the host immune and inflammation responses involved in sepsis and surgery. This study aimed to investigate the potential impact of intraoperative GCs administration on the clinical outcome of surgical patients with abdominal sepsis.

Methods: This retrospective cohort study included a 1:1 propensity score-matched cohort of surgical patients afflicted with abdominal sepsis at 2 medical centers from January, 2008, through December, 2022. Patients were classified into low-GCs, high-GCs, and non-GCs groups according to the dosage of steroids used intraoperatively, and in-hospital mortality was designated as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the Sepsis 3.0 criteria ;
* Patient's age ≥ 18 years;
* Emergency or elective abdominal surgery.

Exclusion Criteria:

* History of severe cardiopulmonary, hepatic, renal, or other organ damage;
* Preoperative presence of infection other than abdominal;
* Unplanned secondary surgery；
* Receiving preoperative glucocorticoid therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abdominal septic patients underwent surgical procedures in two large-scale medical centers (the First Medical Center of the Chinese People's Liberation Army [PLA] General Hospital and the Air Force Medical Center) between Jan, 2008 and Dec, 2022 in Beijing, China.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | January 2008 - December 2022

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, Study Chair — Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital
Locations (1):
- Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital /Depatment of Anesthesiology, The Air Force Medical Center, Beijing, Beijing Municipality, China